CLINICAL TRIAL: NCT03642626
Title: Chimeric Antigen Receptor (CAR)-T Cell Therapy for Patients With Hematologic Malignancies
Brief Title: MT2017-45: CAR-T Cell Therapy for Heme Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS118; MT2017-45 (Other: University of Minnesota Masonic Cancer Center); NCI-2020-04527 (Registry Identifier: CTRP)
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; Large B-cell Lymphoma
Keywords: ALL; CAR-T; CAR19-T; chimeric antigen receptor T cells
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tisagenlecleucel; axicabtagene ciloleucel; fludarabine; Cyclophosphamide; brexucabtagene autoleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- ARM A: Refractory/relapsed B-cell acute lymphoblastic leukemia (ALL) (Experimental)
  Interventions: Drug: KYMRIAH; Drug: Fludarabine 30mg/m2 4 doses; Drug: Cyclophosphamide 500 mg/m2; 2 doses
- ARM B: Yescarta for Refractory diffuse large B cell lymphoma (DLBCL) (Experimental)
  Interventions: Drug: YESCARTA; Drug: Fludarabine 30mg/m2 3 doses; Drug: Cyclophosphamide 500 mg/m2; 3 doses
- ARM C: Kymriah for Refractory diffuse large B cell lymphoma (DLBCL) (Experimental)
  Interventions: Drug: KYMRIAH; Drug: Fludarabine 25mg/m2 3 days; Drug: Cyclophosphamide 250 mg/m2; 3 days
- Arm D: Tecartus CAR-T product for Mantle Cell Leukemia (MCL) (Experimental)
  Interventions: Drug: Fludarabine 30mg/m2 3 doses; Drug: Cyclophosphamide 500 mg/m2; 3 doses; Drug: Tecartus
- Arm E: Breyanzi for relapsed or refractory large B-cell lymphoma (RLBCL) (Experimental)
  Interventions: Drug: Fludarabine 30mg/m2 3 doses; Drug: Cyclophosphamide 500 mg/m2; 3 doses; Drug: Breyanzi Injectable Product
- Arm F: Abecma for relapsed or refractory multiple myeloma (Experimental)
  Interventions: Drug: Fludarabine 30mg/m2 3 doses; Drug: Cyclophosphamide 500 mg/m2; 3 doses; Drug: Abecma, Intravenous Suspension
- Arm G: Tecartus B-cell acute lymphoblastic leukemia (ALL) (Experimental)
  Interventions: Drug: Fludarabine 25mg/m2 3 days; Drug: Tecartus; Drug: Cyclophosphamide 900 mg/m2; 1 day

INTERVENTIONS:
Drug: KYMRIAH — FDA approved CD19-directed genetically modified autologous T cell immunotherapy comprised of autologous T cells
  Other Names: tisagenlecleucel
  Arms: ARM A: Refractory/relapsed B-cell acute lymphoblastic leukemia (ALL); ARM C: Kymriah for Refractory diffuse large B cell lymphoma (DLBCL)
Drug: YESCARTA — CD19-directed genetically modified autologous T cell immunotherapy
  Arms: ARM B: Yescarta for Refractory diffuse large B cell lymphoma (DLBCL)
Drug: Fludarabine 30mg/m2 4 doses — 30 mg/m2 IV daily for 4 doses
  Arms: ARM A: Refractory/relapsed B-cell acute lymphoblastic leukemia (ALL)
Drug: Cyclophosphamide 500 mg/m2; 2 doses — 500 mg/m2 IV daily for 2 doses starting with the first dose of fludarabine
  Arms: ARM A: Refractory/relapsed B-cell acute lymphoblastic leukemia (ALL)
Drug: Fludarabine 30mg/m2 3 doses — 30 mg/m2 IV daily for 3 doses
  Arms: ARM B: Yescarta for Refractory diffuse large B cell lymphoma (DLBCL); Arm D: Tecartus CAR-T product for Mantle Cell Leukemia (MCL); Arm E: Breyanzi for relapsed or refractory large B-cell lymphoma (RLBCL); Arm F: Abecma for relapsed or refractory multiple myeloma
Drug: Cyclophosphamide 500 mg/m2; 3 doses — 500 mg/m2 IV daily for 3 doses starting with the first dose of fludarabine
  Arms: ARM B: Yescarta for Refractory diffuse large B cell lymphoma (DLBCL); Arm D: Tecartus CAR-T product for Mantle Cell Leukemia (MCL); Arm E: Breyanzi for relapsed or refractory large B-cell lymphoma (RLBCL); Arm F: Abecma for relapsed or refractory multiple myeloma
Drug: Fludarabine 25mg/m2 3 days — 25 mg/m2 i.v. daily for 3 days
  Arms: ARM C: Kymriah for Refractory diffuse large B cell lymphoma (DLBCL); Arm G: Tecartus B-cell acute lymphoblastic leukemia (ALL)
Drug: Cyclophosphamide 250 mg/m2; 3 days — 250 mg/m2 IV daily for 3 days starting with the first dose of fludarabine
  Arms: ARM C: Kymriah for Refractory diffuse large B cell lymphoma (DLBCL)
Drug: Tecartus — TECARTUS is a CD19-directed genetically modified autologous T cell immunotherapy, binds to CD19-expressing cancer cells and normal B cells
  Other Names: Brexucabtagene Autoleucel
  Arms: Arm D: Tecartus CAR-T product for Mantle Cell Leukemia (MCL); Arm G: Tecartus B-cell acute lymphoblastic leukemia (ALL)
Drug: Abecma, Intravenous Suspension — Infuse ABECMA 2 days after completion of lymphodepleting chemotherapy.
  Arms: Arm F: Abecma for relapsed or refractory multiple myeloma
Drug: Cyclophosphamide 900 mg/m2; 1 day — Administer cyclophosphamide 900 mg/m2 over 60 minutes on the second day before infusion of TECARTUS
  Arms: Arm G: Tecartus B-cell acute lymphoblastic leukemia (ALL)
Drug: Breyanzi Injectable Product — Infuse BREYANZI 2 to 7 days after completion of lymphodepleting chemotherapy.
  Arms: Arm E: Breyanzi for relapsed or refractory large B-cell lymphoma (RLBCL)

SUMMARY:
This is a phase II study of FDA-approved CAR-T products for patients with hematologic malignancies. Patients will be assigned to Arm A and B based on age and diagnosis. Overall remission rate, safety events and other endpoints will be calculated for Arm A and B separately.

ELIGIBILITY:
ARM A (Kymriah) and Arm G (Tecartus) :Refractory/relapsed B-cell acute lymphoblastic leukemia expressing CD19

Inclusion Criteria:

* Age and Disease Status

  * Must be age 0-25 years (for Arm A Kymriah) or >18 years (Arm G Tecartus)
  * Disease status: Relapsed and refractory pediatric B-cell ALL defined by one of these:

    * Primary induction failure with no complete remission after ≥2 cycles of induction chemotherapy, or
    * Patients with persistent minimal residual disease (MRD >0.01% by flow cytometry or persistent by cytogenetic or molecular assays) after ≥2 cycles of consolidation chemotherapy, or
    * Patients in 2nd or greater relapse of B-ALL or
    * Patients with persistent CNS leukemia, or
    * Down Syndrome or other congenital diseases assuming that they fit the criteria for second or greater relapse or refractory leukemia, or
    * Patients with Ph+ ALL are eligible if theywho have failed or are intolerant to two lines of TKI assuming they fit the criteria for second or greater relapse or are considered refractory.
* Performance Status

  * Arm A: Karnofsky (age ≥16 years) or Lansky (age < 16 years) performance status ≥ 50% at screening; Arm G: ECOG 0, 1 or 2
* Organ Function

  * Renal function defined as:

    * A serum creatinine of ≤1.5 x ULN OR
    * eGFR ≥ 50 mL/min/1.73 m2
  * Liver function defined as:

    ** ALT ≤ 5 times the ULN for age (unless due to disease)

    ** Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
  * Hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram or MUGA
* Other Inclusion Criteria

  * Life expectancy ≥12 weeks
  * Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment.
  * Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Patients with Burkitt's lymphoma/leukemia (i.e. patients with mature B-cell ALL, leukemia with B-cell [sIg positive and kappa or lambda restricted positivity] ALL, with FAB L3 morphology and /or a MYC translocation)
* CNS 2A
* CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to enrollment.
* Patient has taken one of the prohibited concomitant medications within the timeframe outlined in section 6.1

ARM B: Yescarta for Relapsed or Refractory diffuse large B cell lymphoma

Inclusion Criteria:

* Age and Disease Status

  * Adult patients (age ≥ 18 years)Patients must be ≥18 years of age
  * One of the following histologies and expression of CD19 by tumor cells:

    ** diffuse large B-cell lymphoma (DLBCL) not otherwise specified, or

    ** primary mediastinal large B-cell lymphoma, or

    ** high grade B-cell lymphoma, or

    ** DLBCL arising from follicular lymphoma
  * Disease status:

    ** Chemotherapy refractory disease after ≥2 lines of chemotherapy, or

    ** Relapsed with no remission after ≥1 lines of salvage chemotherapy, or

    ** Relapsed following autologous HCT (and failed at least 2 prior lines of therapy including high dose chemotherapy). If salvage therapy is given post autoHCT, the subject must have no response or relapse after the last line of therapy
  * Measurable disease at time of apheresis: Nodal lesions or extranodal lesion
  * ECOG performance status 0-2
  * ALC >/=100/uL at screening (prior to apheresis)
  * Renal function defined as:

    ** A serum creatinine of ≤1.5 x ULN OR

    ** eGFR ≥ 50 mL/min/1.73 m2
  * Liver function defined as:

    * ALT ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
  * Hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram or MUGA
  * Adequate bone marrow reserve (unless marrow infiltrated by disease) defined as :

    * Absolute neutrophil count (ANC) > 1.000/mm3 (only for NHL)
    * Platelets ≥ 50.000/mm3 (transfusion support can be provided)
    * Hemoglobin >8.0 mg/dl (transfusion support can be provided)
  * Life expectancy ≥12 weeks
  * Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment.
  * Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active CNS involvement by malignancy (no evidence of disease in CSF by flow cytometry) CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection (controlled HIV is permissible)
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to apheresis.
* Patient has taken one of the prohibited concomitant medications within the timeframe.

ARM C: Kymriah for rRelapsed or rRefractory diffuse large B cell lymphoma

Inclusion Criteria:

* Age and Disease Status

  * Adult patients (age ≥ 18 years)
  * with relapsed or refractory (r/r) large B-cell lymphoma, including

    * diffuse large B-cell lymphoma (DLBCL) not otherwise specified,
    * high grade B-cell lymphoma
    * and DLBCL arising from follicular lymphoma.
  * Disease status:

    * after two or more lines of systemic therapy or
    * relapse after autologous HCT
* Performance Status

  * ECOG performance status 0-2
  * ALC >/=100/uL at screening (prior to apheresis)
* Organ Function

  * Renal function defined as:

    * A serum creatinine of ≤1.5 x ULN OR
    * eGFR ≥ 50 mL/min/1.73 m^2
  * Liver function defined as:

    * ALT ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
  * Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
  * Hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram or MUGA
  * Adequate bone marrow reserve (unless marrow infiltrated by disease) defined as :

    * Absolute neutrophil count (ANC) > 1.000/mm3 (only for NHL)
    * Platelets ≥ 50.000/mm3 (transfusion support can be provided)
    * Hemoglobin >8.0 mg/dl (transfusion support can be provided)
* Other Inclusion Criteria

  * Life expectancy ≥12 weeks
  * Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment.
  * Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active CNS involvement by malignancy (no evidence of disease in CSF by flow cytometry) CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active or inactive HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to apheresis.
* Patient has taken one of the prohibited concomitant medications within the timeframe

ARM D: Tecartus (Brexucabtagene Autoleucel) for relapsed or refractory mantle cell lymphoma

Inclusion Criteria:

* Age and Disease Status

  * with relapsed or refractory (r/r) mantle cell lymphoma, including
  * prior anthracycline or Bendamustine containing therapy
  * prior Rituximab or other CD20 directed antibody (or inability to treat with CD20 MoAb)
  * not a candidate or relapse after autologous HCT
  * active disease at enrollment
* Performance Status

  *ECOG performance status 0-1
* Organ Function

  * Renal function defined as:

    * A serum creatinine of ≤1.5 x ULN OR
    * eGFR ≥ 50 mL/min/1.73 m2
  * Liver function defined as:

    * ALT ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
* Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
* Hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram or MUGA
* Adequate bone marrow reserve (unless marrow infiltrated by disease) defined as:
* Absolute neutrophil count (ANC) > 1,000/mm^3 (only for NHL)
* Platelets ≥ 50,000/mm^3 (transfusion support can be provided)
* Hemoglobin >8.0 mg/dl (transfusion support can be provided)

Other Inclusion Criteria:

* Life expectancy ≥12 weeks
* Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment. See section 4.5 for definitions of child bearing potential and section 4.6 for definitions of adequate birth control.
* Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active CNS involvement by malignancy (no evidence of disease in CSF by flow cytometry) CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to apheresis (steroids must be stopped >72 hours prior to apheresis).
* Patient has taken one of the prohibited concomitant medications within the timeframe

ARM E: Breyanzi "lisocabtagene maraleucel" for relapsed or refractory large B-cell lymphoma

Inclusion Criteria:

* Age and Disease Status

  * Adult patients (age ≥ 18 years)
  * with relapsed or refractory disease after two or more lines of systemic therapy, including

    * diffuse large B-cell lymphoma (DLBCL) not otherwise specified (including DLBCL arising from indolent lymphoma),
    * high-grade B-cell lymphoma,
    * primary mediastinal large B-cell lymphoma,
    * follicular lymphoma grade 3B
* Performance Status

  *ECOG performance status 0-2
* Organ Function

  * Renal function defined as:

    * A serum creatinine of ≤1.5 x ULN OR
    * eGFR ≥ 30 mL/min/1.73 m2
  * Liver function defined as:

    * ALT ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
* Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
* Hemodynamically stable and LVEF ≥ 40% confirmed by echocardiogram or MUGA
* Adequate bone marrow reserve (unless marrow infiltrated by disease) defined as:

  * Absolute neutrophil count (ANC) > 1,000/mm^3 (only for NHL)
  * Platelets ≥ 50,000/mm^3 (transfusion support can be provided)
  * Hemoglobin >8.0 mg/dl (transfusion support can be provided)

Other Inclusion Criteria:

* Life expectancy ≥12 weeks
* Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment. See section 4.5 for definitions of child bearing potential and section 4.6 for definitions of adequate birth control.
* Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active CNS involvement by malignancy (no evidence of disease in CSF by flow cytometry) CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to apheresis (steroids must be stopped >72 hours prior to apheresis).
* Patient has taken one of the prohibited concomitant medications within the timeframe

ARM F: Abecma "Idecabtagene Vicleucel" for relapsed or refractory multiple myeloma

Inclusion Criteria:

* Age and Disease Status

  * Adult patients (age ≥ 18 years)
  * Relapsed (progression after prior partial or complete remission) or refractory multiple myeloma
  * Evidence of active disease (medullary or extramedullary)
  * Prior therapy (Failure or intolerance to) with an immunomodulatory agent, a proteasome inhibitor, and an antiCD38 monoclonal antibody
* Performance Status

  *ECOG performance status 0-1
* Organ Function

  * Renal function defined as:

    * A serum creatinine of ≤2 x ULN OR
    * eGFR ≥ 50 mL/min/1.73 m2
  * Liver function defined as:

    * ALT ≤ 5 times the ULN for age (unless due to disease)
    * Bilirubin ≤ 2.0 mg/dl with the exception of patients with Gilbert syndrome; may be included if their total bilirubin is ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
* Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation SpO2 > 91% on room air
* Hemodynamically stable and LVEF ≥ 45% confirmed by echocardiogram or MUGA
* Adequate bone marrow reserve (unless marrow infiltrated by disease) defined as:

  * Absolute neutrophil count (ANC) > 1,000/mm^3 (only for NHL)
  * Platelets ≥ 50,000/mm^3 (transfusion support can be provided)
  * Hemoglobin >8.0 mg/dl (transfusion support can be provided)

Other Inclusion Criteria:

* Life expectancy ≥12 weeks
* Women of child bearing potential and sexually active males with partners of child bearing potential must agree to use adequate birth control for the duration of treatment. See section 4.5 for definitions of child bearing potential and section 4.6 for definitions of adequate birth control.
* Written voluntary consent (adults) or parental/guardian consent (minors or adults with diminished capacity) prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy.
* Active CNS involvement by malignancy (no evidence of disease in CSF by flow cytometry) CAR-T is not indicated for the treatment of patients with primary central nervous system lymphoma.
* Presence of Grade 2 to 4 acute or extensive chronic graft-versus-host disease (GVHD). All GVHD medication must be stopped 2 weeks prior to apheresis.
* Uncontrolled active hepatitis B or hepatitis C
* Active HIV infection
* Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to infusion)
* Unstable angina and/or myocardial infarction within 1 month prior to CAR-T infusion
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion
* Intolerance to the excipients of the CAR-T cell product
* Any immunosuppressive medication must be stopped ≥ 2 weeks prior to apheresis (steroids must be stopped >72 hours prior to apheresis).
* Patient has taken one of the prohibited concomitant medications within the timeframe

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2028-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Started | 26 | 44 | 30 | 7 | 13 | 20 | 10
Completed | 26 | 44 | 30 | 7 | 13 | 20 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL) | Total
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 17
  Between 18 and 65 years | 9 | 33 | 14 | 3 | 1 | 6 | 10 | 76
  >=65 years | 0 | 11 | 16 | 4 | 12 | 14 | 0 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 15 | 2 | 4 | 10 | 6 | 58
  Male | 20 | 29 | 15 | 5 | 9 | 10 | 4 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 25 | 43 | 29 | 7 | 11 | 19 | 8 | 142
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  White | 25 | 40 | 26 | 5 | 11 | 18 | 8 | 133
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 3 | 1 | 2 | 0 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 26 | 44 | 30 | 7 | 13 | 20 | 10 | 150

OUTCOME MEASURES:

1. Primary Outcome: Arms B & C&D& E&F: Overall Response Rate (ORR)
Description: ORR defined by complete response + partial response by Lugano
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Arm F: Abecma for Relapsed or Refractory Multiple Myeloma: Fludarabine 30mg/m2 3 doses: 30 mg/m2 IV daily for 3 doses Cyclophosphamide 500 mg/m2; 3 doses: 500 mg/m2 IV daily for 3 doses starting with the first dose of fludarabine Abecma, Intravenous Suspension: Infuse ABECMA 2 days after completion of lymphodepleting chemotherapy.
Arm/Group | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma
Number analyzed (Participants) | 44 | 30 | 7 | 13 | 20
Percentage of participants | 77.3 [63 to 87.2] | 61.3 [43.8 to 76.3] | 100 [59 to 100] | 69.2 [42.4 to 87.3] | 35 [18.1 to 56.7]

2. Primary Outcome: Arm A & E: MRD-negative CR (or CRi)
Description: Percentage of patients with MRD-negative Complete Response CR (or CRi)
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL)
Number analyzed (Participants) | 26 | 13
Percentage of participants | 88.5 [71 to 96] | 100 [75.3 to 100]

3. Secondary Outcome: Percentage of Patients Developing Grade 3 or 4 ICANS
Description: Percentage of patients developing grade 3 or 4 ICANS
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 4 [0 to 21] | 20.5 [11.1 to 34.5] | 3.3 [0 to 17.2] | 42.8 [15.8 to 75] | 0 [0 to 100] | 10 [3.1 to 32.8] | 10 [1.8 to 40.4]

4. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Incidence of treatment related mortality (in absence of disease relapse/progression)
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 0 [0 to 100] | 2.3 [0 to 7] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100]

5. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Incidence of treatment related mortality (in absence of disease relapse/progression)
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 0 [0 to 100] | 2.3 [0 to 7] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100] | 0 [0 to 100]

6. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Incidence of treatment related mortality (in absence of disease relapse/progression)
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 0 [0 to 100] | 7 [0 to 14] | 0 [0 to 100] | 14 [0 to 38] | 15 [0 to 34] | 0 [0 to 100] | 0 [0 to 100]

7. Secondary Outcome: Relapse-free Survival (RFS)
Description: Incidence of Relapse-free Survival (RFS)
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 46 [25 to 68] | 25 [12 to 38] | 47 [28 to 65] | 0 [0 to 100] | 28 [2 to 44] | 55 [35 to 75] | 10 [0 to 28]

8. Secondary Outcome: Event-Free Survival (EFS)
Description: Incidence of event-free survival (EFS) from the date of the CAR-T infusion through 1 year post treatment
Time Frame: 1 Year post treatment
Reporting Status: Not Posted

9. Secondary Outcome: Overall Survival (OS)
Description: Incidence of Overall Survival (OS) from the date of the CAR-T infusion through the date of patient death for any reason.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 26 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 88 [63 to 96] | 86 [72 to 94] | 77 [56 to 88] | 86 [33 to 98] | 69 [37 to 87] | 90 [66 to 97] | 100 [0 to 100]

10. Secondary Outcome: Overall Toxicity
Description: Percentage of patients with grade 3 or 4 targeted toxicity of CRS and/or neurotoxicity
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
Number analyzed (Participants) | 23 | 44 | 30 | 7 | 13 | 20 | 10
Percentage of participants | 21.7 [9.7 to 41.9] | 2.3 [0 to 11.8] | 0 [0 to 100] | 14.3 [2.6 to 51.3] | 0 [0 to 100] | 0 [0 to 100] | 10 [1.8 to 40.4]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL)
All-Cause Mortality (participants affected / at risk) | 0/26 | 3/44 | 0/30 | 1/7 | 2/13 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/44 | 0/30 | 0/7 | 0/13 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/26 | 0/44 | 0/30 | 0/7 | 0/13 | 0/20 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A: Refractory/Relapsed B-cell Acute Lymphoblastic Leukemia (ALL) (N=26) | ARM B: Yescarta for Refractory Diffuse Large B Cell Lymphoma (DLBCL) (N=44) | ARM C: Kymriah for Refractory Diffuse Large B Cell Lymphoma (DLBCL) (N=30) | Arm D: Tecartus CAR-T Product for Mantle Cell Leukemia (MCL) (N=7) | Arm E: Breyanzi for Relapsed or Refractory Large B-cell Lymphoma (RLBCL) (N=13) | Arm F: Abecma for Relapsed or Refractory Multiple Myeloma (N=20) | Arm G: Tecartus B-cell Acute Lymphoblastic Leukemia (ALL) (N=10)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03642626/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03642626/ICF_001.pdf